CLINICAL TRIAL: NCT00102713
Title: An Open Label Study for Treatment of Partial Seizures in Children
Brief Title: A Study for Treatment of Partial Seizures in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M04-714
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Partial Seizures
Keywords: Partial Seizures
MeSH Terms: conditions — Seizures | interventions — Valproic Acid

INTERVENTIONS:
Drug: Divalproex Sodium (Depakote Sprinkle Capsules)

SUMMARY:
The purpose of the study is to assess the safety profile of the investigational medication, Depakote Sprinkle Capsules, in the treatment of partial seizures in children ages 3-10.

ELIGIBILITY:
Inclusion Criteria:

Subject has diagnosis of partial seizures with/without secondary generalization, supported by:

* Observed ictal events consistent with partial seizures with/without secondary generalization; Documented by reliable observers
* 1 of following 3:

  * EEG at some time in past demonstrating focal abnormalities consistent with partial seizures
  * If the EEG is inconclusive or does not support partial seizures, then an MRI/CT will be done
  * If the MRI/CT fails to support a diagnosis of partial seizures, the subject may still qualify based on the principal Investigator's clinical diagnosis
* Subject weighs at least 15 kg (33 lbs).
* Parent/caregiver is able to keep an accurate seizure diary.

Exclusion Criteria:

* Has had status epilepticus in the past 3 months prior to Screening
* Has a history of any of: Cardiac (including clinically important abnormality on ECG); Renal; Psychiatric (including psychosurgery); Oncologic; Endocrine; Metabolic; Pancreatic; Hepatic disease (including clinical/serological history of hepatitis); Urea cycle disorder
* Has: Expanding CNS neoplasm; Active CNS infection; Demyelinating disease; Degenerative neurological disease; Progressive encephalopathy; or any Progressive CNS disease
* Has platelet count less than or equal to 100,000/mcL
* Has blood chemistry ALT/AST value(s) greater than or equal to 2 times upper limit of normal at screening
* Requires anticoagulant drug therapy
* Receiving systemic chemotherapy
* Requires treatment with aspirin
* Subject is pregnant
* Has been on ketogenic diet within 30 days prior to screening
* Considered by investigator to be non-responder to valproate for treatment of epilepsy (e.g., Despite adequate trial with serum concentrations of 60 mcg/mL or greater, subject continues to have inadequate seizure control)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2005-02

PRIMARY OUTCOMES:
Partial Seizure Rate at Week 4

SECONDARY OUTCOMES:
Adverse Events
WASI
WPPSI-III
BASC
UKU-Neurologic Assessment
Vital Signs
Clinical Laboratory Assessments
ECG
PK analysis

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 800-633-9110, Study Director — Abbott
Locations (10):
- United States (10):
  - Neurology Clinic, P.C., Northport, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Child Neurology Associates, P.C., Atlanta, Georgia
  - Akron Children's Hospital, Akron, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Texas Association of Pediatric Neurology, P.A., San Antonio, Texas
  - Monarch Medical Research, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Richard V. Colan, M.D., S.C., Milwaukee, Wisconsin